CLINICAL TRIAL: NCT04936230
Title: Phase II Randomized Trial of Immunotherapy Versus Immunotherapy and Radiation Therapy for Platinum Ineligible/Refractory Metastatic Urothelial Cancer (IMMORTAL)
Brief Title: Immunotherapy With or Without Radiation Therapy for Metastatic Urothelial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-06326; NCI-2021-06326 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A032002 (Other: Alliance for Clinical Trials in Oncology); A032002 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2021-06-22; First posted 2021-06-23 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Urothelial Carcinoma; Platinum-Resistant Urothelial Carcinoma; Stage IV Bladder Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 25-40 minutes on day 1 of each cycle. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, bone scan and/or PET scan, as well as optional urine and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Arm B (pembrolizumab, SBRT) (Experimental): Patients receive pembrolizumab as in Arm A. Patients also undergo SBRT QD every other day for 3 fractions over 2 weeks that must be completed before 12 weeks after the first dose of pembrolizumab in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, bone scan, and/or PET scan, as well as optional urine and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; QL2107; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Arm B (pembrolizumab, SBRT)

SUMMARY:
This phase II trial compares the effect of adding radiation therapy to an immunotherapy drug called pembrolizumab versus pembrolizumab alone in treating patients with urothelial cancer that has spread from where it first started (primary site) to other places in the body (metastatic). The addition of radiation to immunotherapy may shrink the cancer, but it could also cause side effects. Immunotherapy with monoclonal antibodies such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Stereotactic body radiation therapy (SBRT) is a type of radiation therapy that uses high energy x-rays to kill tumor cells and shrink tumors. This method uses special equipment to position a patient and precisely deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and may cause less damage to normal tissue than conventional radiation therapy. The combination of pembrolizumab and radiation therapy may be more efficient in killing tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the overall response rates by 6 months in patients with advanced urothelial carcinoma when treated with immunotherapy alone and immunotherapy plus radiotherapy to a single site.

SECONDARY OBJECTIVES:

I. To compare the response rates using immune related Response Evaluation Criteria in Solid Tumors (iRECIST) as assessed by central review.

II. To compare progression-free survival (PFS) and overall survival (OS) for patients treated with immunotherapy and immunotherapy plus radiotherapy.

III. To compare the rates of treatment discontinuation at 1 year. IV. To assess adverse events experienced by patients treated with immunotherapy and immunotherapy plus radiotherapy via the Common Terminology Criteria for Adverse Events (CTCAE) and Patient Reported Outcome (PRO)-CTCAE.

IV. To determine whether treatment effects are similar for key subgroups including those defined by the stratification variables.

QUALITY OF LIFE CORRELATIVE STUDY OBJECTIVES:

I. To compare patient-reported fatigue as assessed by the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue 8a from baseline through 24 months between patients treated with immunotherapy alone and immunotherapy plus radiotherapy to a single site.

II. To compare health-related quality of life (HRQOL) as assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Core (C)30 from baseline through 24 months between patients treated with immunotherapy alone and immunotherapy plus radiotherapy to a single site.

III. To compare urinary symptoms as assessed by the EORTC QLQ-BLM30 from baseline through 24 months between patients treated with immunotherapy alone and immunotherapy plus radiotherapy to a single site.

IV. To compare patient-reported diarrhea, shortness of breath and pain as assessed by the EORTC QLQ-C30 from baseline through 24 months between patients treated with immunotherapy alone and immunotherapy plus radiotherapy to a single site.

V. To compare health utilities and quality-adjusted survival between patients treated with immunotherapy alone and immunotherapy plus radiotherapy to a single site.

VI. To compare other scale scores of the EORTC QLQ-C30 (global health status and quality of life; physical, role, emotional, cognitive, and social function; symptoms) and EORTC QLQ-BLM30 (urostomy problems, catheter problems, future perspectives, abdominal bloating and flatulence, body image, sexual function) at 45 days, and at 6, 12, and 24 months between patients treated with immunotherapy alone and immunotherapy plus radiotherapy to a single site.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive pembrolizumab intravenously (IV) over 25-40 minutes on day 1 of each cycle. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan, magnetic resonance imaging (MRI), bone scan and/or positron emission tomography (PET) scan, as well as optional urine and blood sample collection throughout the study.

ARM B: Patients receive pembrolizumab as in Arm A. Patients also undergo SBRT once daily (QD) every other day for 3 fractions over 2 weeks that must be completed before 12 weeks after the first dose of pembrolizumab in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, bone scan, and/or PET scan, as well as optional urine and blood sample collection throughout the study.

After completion of study treatment, patients are followed up within 12 weeks and then every 3 months for 3 years following registration.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic urothelial carcinoma
* Patients must be either ineligible for platinum treatment or platinum refractory as defined below:

  * Platinum-ineligible: If patients meet any one of the following criteria:

    * Impaired renal function (creatinine clearance [CrCl] of < 30 mL/min)
    * Eastern Cooperative Oncology Group (ECOG) performance status (PS) of > 2
    * Grade > 2 peripheral neuropathy
    * New York Heart Association (NYHA) Heart Failure of > 3
  * Platinum-refractory: If patients meet any one of the following criteria:

    * Prior platinum-based perioperative chemotherapy within 12 months of relapse
    * Prior platinum-based chemotherapy for metastatic disease
* Patients must have at least one measurable site >= 1 cm in diameter per RECIST 1.1 and a site targetable for radiotherapy. Measurable site must not overlap with radiated site such that measurable site cannot receive > 2 Gy per fraction
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions)
* Men and women, ages >= 18 years of age
* ECOG performance status =< 2
* Leukocytes >= 2,500/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 8 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x upper limit of normal (ULN)

  * AST and/or ALT =< 5 x ULN for patients with liver involvement
* Alkaline phosphatase =< 2.5 x ULN

  * =< 5 x ULN for patients with documented liver involvement or if due to bone metastases primarily in absence of liver disease, no limitation
* No prior allogeneic bone marrow transplantation or prior solid organ transplantation
* No prior radiotherapy to targetable site or measurable site
* No chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events (other than alopecia) due to agents administered more than 4 weeks earlier. However, the following therapies are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Palliative radiotherapy for bone metastases > 2 weeks prior to registration
* No prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* No treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* No prior treatment with any other investigational agent within 4 weeks prior to registration
* No prior treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 6 weeks prior to registration
* Any prior systemic therapy is permitted except therapy with PD1/PDL1 inhibitor
* Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
* The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* No active tuberculosis (TB)
* No known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Patients with known primary central nervous system (CNS) malignancy or symptomatic CNS metastases are excluded, with the following exceptions:

  * Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

    * Evaluable or measurable disease outside the CNS
    * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
    * No history of intracranial hemorrhage or spinal cord hemorrhage
    * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted
    * No neurosurgical resection or brain biopsy within 28 days prior to registration
* Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

  * Radiographic demonstration of improvement upon the completion of CNS directed therapy and no evidence of interim progression between the completion of CNS directed therapy and the screening radiographic study
  * No stereotactic radiation or whole-brain radiation within 28 days prior to registration
  * Screening CNS radiographic study >= 4 weeks from completion of radiotherapy and >= 2 weeks from discontinuation of corticosteroids
* No active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible
* No known history of, or any evidence of active, non-infectious pneumonitis or colitis
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* No known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; or inherited liver disease causing decompensated cirrhosis
* No history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* No significant cardiovascular disease (such as New York Heart Association class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* No other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* No history of leptomeningeal disease
* No uncontrolled tumor-related pain
* Patients requiring pain medication must be on a stable regimen at study entry
* Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period
* Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment
* No uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

  * Patients with indwelling catheters (e.g., PleurX [registered trademark]) are allowed
* Patients with controlled type 1 diabetes mellitus on a stable insulin regimen are eligible
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

  * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
  * Rash must cover less than 10% of body surface area (BSA)
  * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
* No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No active infections requiring systemic antibiotics within 2 weeks prior to registration. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* No major surgical procedure within 28 days prior to registration or anticipation of need for a major surgical procedure during the course of the study
* No administration of a live, attenuated vaccine within 30 days before registration or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of immunotherapy
* Patients who have received live attenuated vaccines within 30 days of the first dose of trial treatment are eligible at the discretion of the investigator. All seasonal influenza vaccines and vaccines intended to prevent severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease 2019 (COVID-19) are allowed
* Physicians should consider whether any of the following may render the patient inappropriate for this protocol:

  * Patients with life expectancy of less than 6 months
  * Psychiatric illness which would prevent the patient from giving informed consent
  * Medical conditions such as uncontrolled infection, uncontrolled diabetes mellitus or cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient

    * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
    * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
    * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
  * Patients with a "currently active" second malignancy other than non-melanoma skin cancers or cervical carcinoma in situ. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for >= 3 years
* Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study and for 4 months (120 days) after the last dose of study agent due to the teratogenic potential of the therapy utilized in this trial. Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives or double barrier method (diaphragm plus condom). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Himanshu Nagar, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (83):
- United States (83):
  - Littleton Adventist Hospital, Littleton, Colorado
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - NYP/Weill Cornell Medical Center, New York, New York
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - VCU Massey Cancer Center at Hanover Medical Park, Mechanicsville, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Pembrolizumab) | Arm B (Pembrolizumab, SBRT)
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: In order to maintain the deidentification of the 1 patient accrued, the patient demographics will not be shared.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Pembrolizumab) | Arm B (Pembrolizumab, SBRT) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Will be defined as a complete response (CR) or partial response (PR) as assessed by the treating physician using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
Time Frame: Up to 6 months from randomization
Population: In order to maintain the deidentification of the 1 patient accrued, this outcome measure will not be shared.
Arm/Group | Arm A (Pembrolizumab) | Arm B (Pembrolizumab, SBRT)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Tumor Response
Description: Will be determined to have a tumor response if they have a CR or PR as assessed by immune modified RECIST.
Time Frame: Up to 3 years from randomization
Population: In order to maintain the deidentification of the 1 patient accrued, this outcome measure will not be shared.
Arm/Group | Arm A (Pembrolizumab) | Arm B (Pembrolizumab, SBRT)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Stratified Cox models will be used to compare the outcomes between the two treatment groups. The results will be summarized with a forest plot displaying the estimate of the hazard ratio and corresponding 95% confidence interval.
Time Frame: Time from randomization until disease progression as assessed by the treating physician using RECIST 1.1 or death due to any cause, assessed up to 3 years
Population: In order to maintain the deidentification of the 1 patient accrued, this outcome measure will not be shared.
Arm/Group | Arm A (Pembrolizumab) | Arm B (Pembrolizumab, SBRT)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival
Description: as for outcome 3
Time Frame: Time from randomization until death due to any cause. Patients who are not known to be dead at time of analysis will be censored at the time of their last follow-up, assessed up to 3 years
Population: In order to maintain the deidentification of the 1 patient accrued, this outcome measure will not be shared.
Arm/Group | Arm A (Pembrolizumab) | Arm B (Pembrolizumab, SBRT)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Rate of Treatment Discontinuation
Description: The proportion of patients who discontinue their protocol directed treatment prior to one year from date of study registration will be determined. Patients who stop their protocol directed treatment for any reason prior to one year from study registration will be considered to have discontinued their treatment. The rates of treatment discontinuation at one year will be summarized with a binomial point estimate and corresponding 95% confidence interval by arm. A comparison between the rates will be performed with a chi-square test or a Fisher's exact test if the assumptions of the chi-square test are violated.
Time Frame: At 1 year
Population: In order to maintain the deidentification of the 1 patient accrued, this outcome measure will not be shared.
Arm/Group | Arm A (Pembrolizumab) | Arm B (Pembrolizumab, SBRT)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Incidence of Adverse Events
Description: Will be assessed by Common Terminology Criteria for Adverse Events version 5.0. Adverse events will be summarized with frequencies and relative frequencies.
Time Frame: Up to 3 years from randomization
Population: In order to maintain the deidentification of the 1 patient accrued, this outcome measure will not be shared.
Arm/Group | Arm A (Pembrolizumab) | Arm B (Pembrolizumab, SBRT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: In order to maintain the deidentification of the 1 patient accrued, this outcome measure will not be shared.
Arm/Group | Arm A (Pembrolizumab) | Arm B (Pembrolizumab, SBRT)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT04936230/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT04936230/ICF_001.pdf